CLINICAL TRIAL: NCT04653649
Title: Immunotherapy With Autologous CAR30 T Cells for Patients With Classic Hodgkin Lymphoma and Non-Hodgkin T-cell Lymphoma With CD30 Expression.
Brief Title: CAR T-cells Against CD30 (HSP-CAR30) for Relapsed/ Refractory Hodgkin and T-cell Lymphoma.
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Josep Carreras Leukaemia Research Institute (Other); Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIBSP-CAR-2019-30
Record Dates: First submitted 2020-11-18; First posted 2020-12-04 (Actual); Last update posted 2020-12-04 (Actual); Status verified 2020-11

CONDITIONS: Hodgkin Lymphoma, Adult; T Cell Lymphoma
MeSH Terms: conditions — Hodgkin Disease; Lymphoma, T-Cell

STUDY DESIGN:
Intervention Model Description: Experimental: HSP-CAR30 (anti-CD30 CAR T cells)
  Dose escalation phase:
  Phase I:
  Ten patients will be treated with HSP-CAR30 (anti-CD30 CAR T-cells) with an escalation approach to define maximum tolerated dose (MTD) from 3 x 106/kg to 10 x 106/kg.
  Phase IIa:
  Twenty patients will be treated with HSP-CAR30 at MTD to evaluate efficacy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HSP-CAR30 (anti-CD30 CAR T cells) (Experimental): Phase I:
  Ten patients will be treated with HSP-CAR30 (anti-CD30 CAR T-cells) with an escalation approach to define maximum tolerated dose (MTD) from 3 x 106/kg to 10 x 106/kg.
  Phase IIa:
  Twenty patients will be treated with HSP-CAR30 at MTD to evaluate efficacy.
  Interventions: Biological: HSP-CAR30

INTERVENTIONS:
Biological: HSP-CAR30 — Anti-CD30 CAR T-cells

SUMMARY:
HSP-CAR30 is a cell suspension of genetically modified T-cells to express a second generation (4-1BBz) chimeric antigen receptor (CAR) directed against CD30.

This is a phase I/IIa, interventional, single arm, open label, treatment study to evaluate the safety, tolerability and efficacy of HSP-CAR30 in patients with relapsed/refractory Hodgkin lymphoma and relapsed/refractory T-cell lymphoma expressing CD30.

ELIGIBILITY:
Inclusion Criteria:

* Classic Hodgkin lymphoma:

  * Relapsed patients after autologous hematopoietic stem cell transplantation who have already received Brentuximab-Vedotin and anti-PDL1 antibodies, OR
  * Primarily refractory patients who do not reach CR after rescue, including Brentuximab-Vedotin and anti-PDL1 antibodies.
* Anaplastic large T-cell lymphoma (ALK+/ALK-) and peripheral T-cell lymphoma (NOS/Angioimmunoblastic):

  * >90% of tumor cells expressing CD30 determined by immunohistochemistry, AND
  * Relapsed patients after autologous hematopoietic stem cell transplantation, OR
  * Primarily refractory patients (after first line, including anthracycline) who do not achieve CR after rescue.
  * All patients must sign an informed consent before starting any procedure.
  * All patients must have measurable disease (detected by PET-CT) at the time of inclusion.
  * Performance status: ECOG 0-1
  * FEV1> 39%; DLCO and FVC> 39% of NV.
  * No significant ventricular dysfunction: EF >45%.
  * Total bilirubin and transaminases <3 times the maximum normal value, unless attributable to lymphoma.
  * Creatinine <2 times the normal maximum value and clearance> 40 mL/min.

Exclusion Criteria:

* Performance status: ECOG 2-4
* Prior allogeneic haematopoietic stem cell transplant.
* Active hepatitis B, C or HIV infection
* Active bacterial, fungal, or viral infection.
* Evidence of CNS involvement by lymphoma.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-29 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
To assess safety and toxicity of the administration of autologous anti-CD30 CAR T-cells | 12 months
  Number of patients with cytokine release syndrome and/or ICANs grade 1-4 according to ASBMT Consensus
To establish the maximum tolerated dose (MTD; defined as the dose that induces maximum limiting toxicity) of autologous anti-CD30 CAR T-cells in patients with refractory or relapsed classic Hodgkin or CD30 + T NHL. | 12 months
  Number of patients receiving maximum dose (1 x 10e7/kg CART+ cells) without DLT
To analyze the rate of complete responses at 3 months after the procedure | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Santa Creu i Sant Pau, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caballero AC, Ujaldon-Miro C, Pujol-Fernandez P, Montserrat-Torres R, Guardiola-Perello M, Escudero-Lopez E, Garcia-Cadenas I, Esquirol A, Martino R, Jara-Bustamante P, Ezquerra P, Soria JM, Iranzo E, Moreno-Martinez ME, Riba M, Sierra J, Alvarez-Fernandez C, Escriba-Garcia L, Briones J. HSP-CAR30 with a high proportion of less-differentiated T cells promotes durable responses in refractory CD30+ lymphoma. Blood. 2025 Apr 17;145(16):1788-1801. doi: 10.1182/blood.2024026758. PMID 39841453